CLINICAL TRIAL: NCT01687439
Title: Effect of Endostar Combined With Chemotherapy and Radiotherapy on Blood Vessels and Microenvironment of Tumor for Non-small Cell Lung Cancer
Brief Title: Effect of Endostar Combined With Chemotherapy and Radiotherapy on Blood Vessels and Microenvironment of Tumor for Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Fan Ming, Associate Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSCLC0901
Record Dates: First submitted 2012-08-16; First posted 2012-09-19 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-09

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — endostar protein; Vinorelbine; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Eligible patients receive one cycle of Endostar monotherapy, two cycles of Endostar combined with chemotherapy (vinorelbine plus cisplatin) treatment, followed by Endostar plus radiotherapy treatment.
  Interventions: Drug: Endostar; Drug: Vinorelbine; Drug: Cisplatin; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Endostar — 7.5mg/m2, D1-14
Drug: Vinorelbine — 25-30mg/m2, D1,8
Drug: Cisplatin — 25 mg/m2, D1-3
Radiation: Radiotherapy

SUMMARY:
Primary objective: functional imaging and quantitative imaging detection of the effects of Endostar combined with chemotherapy and radiotherapy on Non-small Cell Lung Cancer (NSCLC).

Secondary objective: To evaluate 1) the role of Endostar in regulating tumor vessels and normalizing of microenvironment; 2) Toxicity of Endostar combined with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven inoperable stage IIIb-IV NSCLC
* ECOG PS 0-1
* Life expectancy > 3 months
* Adequate blood functions: Absolute neutrophil count (ANC) ≥ 1.5 x 109/L, platelet count ≥ 100 x 109/L, and hemoglobin ≥ 9 g / dL
* Adequate liver function: total bilirubin <1.5 times the upper limit of normal (ULN); AST and ALT <2.5 times ULN in patients without liver metastases, <5 times ULN in patients with liver metastases
* Adequate renal function: serum creatinine ≤ 1.25 times ULN or calculated creatinine clearance ≥ 50 mL / min and urinary protein <2+. In patients with baseline urinary protein ≥ 2+, 24 hours urine should be collected and 24 hours urine protein ≤ 1g
* International normalized ratio (INR) ≤ 1.5 and prothrombin time(PT) ≤ 1.5 times ULN within 7 days before enrollment
* Written informed consent

Exclusion Criteria:

* Evidence of bleeding diathesis or coagulopathy
* History of hemoptysis, defined as bright red blood more than half a teaspoon 3 months before enrollment
* Previously received chemotherapy and radiotherapy and biological targeted therapy
* Uncontrolled hypertension (systolic blood pressure> 150 mmHg and/or diastolic blood pressure> 100 mm Hg)
* Clinically significant (ie, active) cardiovascular diseases, such as cerebrovascular accident (within 6 months before initiating treatment), myocardial infarction (within 6 months before initiating treatment), unstable angina, congestive heart failure (New York Heart Association class ≥Grade II) , serious arrhythmia which needs medication during the study and may affect the study or can not be controlled by drugs
* Unhealed wounds, active peptic ulcer or fracture
* Gastrointestinal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months before enrollment
* Women with intact uterus (menopause more than two years excluded) who are unwilling to take effective non-hormonal contraception (IUD, spermicide barrier birth control device or sterilization) during the study. Male who are unwilling to take effective contraceptive measures during the study
* Participated in other clinical trials within 28 days before the initiation of treatment.
* Allergic to any of the study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-12; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Tumor blood volume | 3 months
Tumor blood flow | 3 months
Permeability-surface area product | 3 months
18-FDG PET SUV values | 3 months

SECONDARY OUTCOMES:
The incidence of adverse events | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Guoliang Jiang, MD, Principal Investigator — Fudan University; Ming Fan, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China